CLINICAL TRIAL: NCT03118661
Title: Effect of CCR5 Inhibition by Maraviroc on HIV-1 Infected Subjects Who Require Allogeneic Hematopoietic Cell Transplant for Any Indication and Its Observed Effect on Graft Versus Host Disease and HIV-1 Persistence
Brief Title: Maraviroc on HIV-1 Infected Subjects Who Require Allogeneic Hematopoietic Cell Transplant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No accrual to the study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201704019
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maraviroc after allo-HCT (Experimental): * Step 1: participants who have received at least 30 days of maraviroc immediately post allo-HCT can be enrolled. Blood will be drawn at 2 time points at least 2 weeks apart, but within 4 weeks, and assessed for HIV-1 reservoir using both DNA assays and cell-associated reactivation by infectivity after stimulation. If any biopsies post allo-HCT are performed as part of standard of care and available, these will also be assessed for HIV-1
  * Step 2: If HIV-1 reservoir is undetecable, antiretrovirals (ART) will be stopped in a structured treatment interruption (STI). HIV-1 VLs and CD4+ T-cells check weekly. Week 16, participants will have a large volume blood draw if remain suppressed. If confirmed return of viremia, ART will be reinitiated and he/she will be followed until HIV VL is <50 copies/ml. If he/she remains suppressed at Week 16 and repeat assays confirm no detectable HIV-1, HIV-1 VLs and CD4+ T-cell counts will be checked monthly until Week 52, and then quarterly until Year 5
  Interventions: Other: For Step 2: Structured treatment interruption; Procedure: Peripheral blood draw

INTERVENTIONS:
Other: For Step 2: Structured treatment interruption — -Accepted tool in the evaluation of immunological interventions, gene therapy, or therapeutic vaccines for the treatment of HIV infection
  Other Names: STI
Procedure: Peripheral blood draw — -Screening, entry for Step 1, Step 1 visit 2, entry for Step 2, weekly, week 16, monthly through week 52, week 52, quarterly through year 5, year 5, and viral relapse

SUMMARY:
The goal of this proposal is to determine the effect of maraviroc when it has been a part of the antiretroviral (ART) regimen given immediately after allogeneic hematopoietic cell transplant (allo-HCT) for HIV-1 infected participants who have a hematopoietic malignancy or other underlying disorder requiring an allogeneic transplant. Maraviroc has been given in practice to alleviate symptoms of graft vs. host disease (GvHD). Given its mechanism of action, it may also have an effect on the reservoir size of HIV-1 in infected patients. This study will inform potential future studies, evaluating the effect of this approach on the incidence and severity of GvHD, and determining its effect on HIV-1 reservoir.

ELIGIBILITY:
Inclusion Criteria (Step 1)

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA VL.
* Receipt of allo-HCT for any indication at least 100 days prior to study entry.
* Receipt of maraviroc for at least 30 days starting at date of transplant. Longer receipt of maraviroc is acceptable. Documentation of HIV-1 tropism for CCR5 should be obtained if available, but it is not necessary that the participant have prior CCR5-tropic.
* At least 18 years of age.
* HIV-1 RNA that is <50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 45 days prior to study entry.
* For females of reproductive potential (i.e., women who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative urine pregnancy test (with a sensitivity of 15-25 mIU/mL) within 48 hours prior to screening and entry.
* Negative HBsAg result obtained within 6 months prior to study entry, or documentation of HBV immunity by positive HBV sAb at any time
* The following laboratory values obtained within 45 days prior to enrollment:

  * CD4+ T cell count >250 cells/ mm^3
  * Absolute neutrophil count (ANC) ≥1000 cells/mm^3
  * Hemoglobin ≥10.0 g/dL for men and ≥9.0 g/dL for women
  * Platelet count ≥ 50,000/mm3
* Ability and willingness of participant or legal representative to provide informed consent.

Additional Inclusion Criteria for Step 2 of Study:

* HIV-1 latent reservoir undetectable by co-culture and DNA
* No confirmed detectable HIV-1 RNA > 1000 cells/mm3 since discontinuation of maraviroc
* Prior HIV-1 genotype results that confirm that there are active agents available in at least three classes of ART drugs (NRTI, NNRTI, PI or integrase).
* Willing to stop ART
* Willing to undergo high volume blood draw (125 cc) at Week 16
* Willing to restart ART if HIV-1 viremia returns
* Provide informed consent for Step 2

Exclusion Criteria:

* Ongoing AIDS-related opportunistic infection (including oral thrush).
* Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
HIV-1 proviral DNA levels in peripheral blood | Up to week 16 after transplant
  * Obtained from peripheral blood
  * Used to determine if participant can proceed to Step 2
HIV-1 reactivation in stimulated assay | Up to week 16 after transplant
  * Obtained from peripheral blood
  * Used to determine if participant can proceed to Step 2
Presence and severity of GvHD | Through 5 years after transplant
  -GvHD will be measured using the NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-Versus-Host Disease: IV. Response Criteria Working Group Report
Time to hematopoietic cell and immune recovery | Up to 100 days after transplant
  -In general, the mean time of engraftment of the donor cells is approximately 90 to 100 days post-transplant and this can be monitored by measuring the percent chimerism of donor cells.
Number of participants who experience chimerism | At the time of screening
  -Chimerism is measured by ≥ 98% of blood cells donor derived
Survival of participants | 100 days after transplant
  -Number of participants who are alive 100 days after transplant
Survival of participants | Week 26 after transplant
  -Number of participants who are alive 26 weeks after transplant
Survival of participants | Week 52 after transplant
  -Number of participants who are alive 52 weeks after transplant
Survival of participants | 5 years after transplant
  -Number of participants who are alive 5 years after transplant
Event free survival | 100 days after transplant
  -Defined as survival where the cancer does not recur, the graft takes, and there are no life-threatening events
Event free survival | Week 26 after transplant
  -Defined as survival where the cancer does not recur, the graft takes, and there are no life-threatening events
Event free survival | Week 52 after transplant
  -Defined as survival where the cancer does not recur, the graft takes, and there are no life-threatening events
Event free survival | 5 years after transplant
  -Defined as survival where the cancer does not recur, the graft takes, and there are no life-threatening events

SECONDARY OUTCOMES:
Number of participants who achieve a state of functional cure | Through 5 years after transplant
  -Functional Cure: Following the discontinuation of all HIV-1 related treatment interventions, including HAART, a participant will be considered to have achieved an HIV-1 functional cure if for at least 5 years they: maintain an undetectable plasma viral load, using standard clinical assays, have achieved full CD4+ lymphocyte recovery with normal levels of T cell activation and proliferation, and normal levels of immunoglobulins with no disease progression. It is anticipated that participants who have achieved a functional cure will continue to have detectable HIV-1 DNA in peripheral blood cells and/or tissues.
Number of participants who achieve a state of sterilizing cure | Through 5 years after transplant
  -Sterilizing cure: same definition of functional cure but no detectable replication-competent virus in peripheral blood and minimal (near limits of detection) HIV-1 DNA in peripheral blood and or tissue
Number of participants who have plasma viral load <50 copies/ml | Through 5 years after transplant
  -Obtained from peripheral blood
Number of participants who have existence of replication competent HIV-1 reservoirs in peripheral blood, gut and other tissue compartments | Through 5 years after transplant
  -Obtained from peripheral blood
Number of participants who have gut immune reconstitution | Through 5 years after transplant
  -Will consist of tissue immunohistochemistry to analyze CD4 T cells when feasible, and for plasma markers of gut microbial translocation namely lipopolysaccharide (LPS) and soluble CD14 (sCD14) a marker of monocyte activation attributed to LPS effects

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Presti, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu